CLINICAL TRIAL: NCT06965062
Title: Cervical Lymphatico-Venous Bypass for Treatment of Alzheimer's Disease - Proof of Concept Study (CLyVeB-AD-1 Study)
Acronym: CLyVeB-AD-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vincent Tay Khwee Soon (Other)
Collaborators: Changi General Hospital (Other); Singapore General Hospital (Other); National Neuroscience Institute (Other)
Responsible Party: Sponsor-Investigator, Vincent Tay Khwee Soon, Consultant Plastic Surgeon, Changi General Hospital
Organization: Changi General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ClyVeB-AD-1
Record Dates: First submitted 2025-01-17; First posted 2025-05-11 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease; Dementia Alzheimer Type; Dementia Alzheimer's Type; Alzheimer's Disease; Alzheimer's Disease (AD)
Keywords: Alzheimer's Disease; Dementia; lymphatic surgery; lymphaticovenous anastomosis; lymphaticovenous bypass; cervical lymph node; meningeal lymphatic system; glymphatic system
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical Intervention (Experimental): This is single-arm, open-label proof of concept study.
  Interventions: Procedure: Deep cervical lymph node to venous bypass (DCLNV-BP)

INTERVENTIONS:
Procedure: Deep cervical lymph node to venous bypass (DCLNV-BP) — Participants will under bilateral deep cervical lymph node to venous bypass procedure under general anaesthesia.
  Other Names: Lymphaticovenous anastomosis

SUMMARY:
Alzheimer's disease (AD), one of the most common causes of dementia in Singapore and the developed world, is a neurodegenerative disorder with high socioeconomic impact. Accumulation of neurotoxic proteins (ie. amyloid, tau) are purported to lead to neuroinflammation, synaptic dysfunction and cognitive decline. The available pharmacotherapy provide limited symptomatic control, modest effect on disease progression with significant risk of side effects. Patients with AD eventually run out of effective pharmacotherapy and deteriorate.

Recent evidence implicated the glymphatic system, meningeal lymphatics of the brain, and downstream drainage to the cervical lymphatic system in the accumulation of neurotoxic proteins in AD. This presented the opportunity for extra-cranial intervention, and has since been demonstrated in preclinical models. Based on these development, Xie and colleagues pioneered the deep cervical lymph node to venous bypass (DCLNV-BP) procedure with very promising early outcomes. The observed improvement had been attributed to enhanced clearance of the neurotoxic proteins. Knowledge gap and clinical equipoise remain, and clinical trials are required to understand the safety, mechanism of action, patient selection, and long-term outcomes.

In this proof of concept study, the investigators aim to assess safety and preliminary efficacy of DCLNV-BP in AD. An approach using objective clinical assessments, biomarkers and neuroimaging, to assess safety, evaluate preliminary efficacy and elucidate the possible mechanism underlying the observed effects, is undertaken. Since there are limited effective treatment for AD, this procedure is potentially ground breaking if it proves to halt progression or even improve patients' cognition, function and behaviour. Indirectly, this will have enormous health economic benefit for Singapore and the developed world that is facing the silver tsunami. Findings from this pilot study will lay the groundwork for future trials and research collaboration in AD and other neurodegenerative diseases.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild-moderate Alzheimer's disease (based on NIA-AA criteria);
* Mini-Mental State Examination (MMSE) score 10-22;
* Both participants and caregiver are able to understand English or Mandarin
* Ability to provide informed consent or have a legally authorised representative to provide informed consent;
* Good family support for post-treatment care and rehabilitation;
* Fit for general anaesthesia/deep sedation and surgery (ASA 1-2; excluding the diagnosis of Alzheimer's Disease).

Exclusion Criteria:

* Cognitive decline due to prior infection or autoimmune diseases;
* History of major cerebrovascular events or significant cardiovascular diseases;
* Inability to have the head turned passively by at least 40 degrees;
* Previous neck lymph node surgery or irradiation;
* Active infection or malignancy;
* Any contraindications to surgery or lumbar puncture
* Any contraindication to MRI/PET scan (eg. metallic implant that are not MRI-safe, known radiotracer allergy)
* Experimental Alzheimer's Disease treatment within the past 6 months. • Current use of monoclonal antibodies treatment (eg. lecanemab/donanemab)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety: Number of treatment-related adverse events | Over 2 years
  Treatment related adverse events and postoperative side effects eg. anaesthetic complications, infection, seroma, nerve or vascular injuries, wound healing issues, death.
Mini Mental State Examination | Over 2 years
  Quick assessment of the cognitive domain. Assessment to be performed at: (1) Baseline; (2) Postoperative(PO) day 3; (3) PO day 7; (4) PO day 14; (5) PO 6 week; (6) PO 3 months; (7) PO 6 months; (8) PO 1 year; (9) PO 2 years.
Montreal Cognitive Assessment | Over 2 years
  Brief assessment of the cognitive domains, especially in mild cognitive impairment, for memory, visuospatial skills, executive function. Assessment to be performed at: (1) Baseline; (2) Postoperative(PO) day 14; (3) PO 6 week; (4) PO 3 months; (5) PO 6 months; (6) PO 1 year; (7) PO 2 years.
Clinical Dementia Rating (CDR) | Over 2 years
  Assessment administered to the participant and caregiver to test various cognitive domains (ie. orientation, attention and working memory, memory, visuospatial, language, executive function) and activities of daily living. Assessment to be performed at: (1) Baseline; (2) Postoperative(PO) day 14; (3) PO 6 week; (4) PO 3 months; (5) PO 6 months; (6) PO 1 year; (7) PO 2 years.
Neuropsychiatric Inventory (NPI) | Over 2 years
  A comprehensive assessment of neuropsychiatric symptoms in patients with dementia, specifically behavioral changes, and administered to the main caregiver over about 5 minutes. Assessment to be performed at: (1) Baseline; (2) Postoperative(PO) day 14; (3) PO 6 week; (4) PO 3 months; (5) PO 6 months; (6) PO 1 year; (7) PO 2 years.
Geriatric Depression Scale-Short Form (GDS-SF) | Over 2 years
  This assessment will take 5-7 minutes and will be administered to the participant to measure depressive symptoms. Assessment to be performed at: (1) Baseline; (2) Postoperative(PO) day 14; (3) PO 6 week; (4) PO 3 months; (5) PO 6 months; (6) PO 1 year; (7) PO 2 years.
Quality of Life - Alzheimer's Disease (QoL-AD) | Over 2 years
  This assessment will take 5-10 minutes and will be administered to the participant to measure Quality of Life measures in AD. Assessment to be performed at: (1) Baseline; (2) Postoperative(PO) day 14; (3) PO 6 week; (4) PO 3 months; (5) PO 6 months; (6) PO 1 year; (7) PO 2 years.
Zarit Burden Score | Over 2 years
  This assessment will take take 5-10 minutes and will be administered to the main caregiver to ascertain changes in caregiver burden.. Assessment to be performed at: (1) Baseline; (2) Postoperative(PO) day 14; (3) PO 6 week; (4) PO 3 months; (5) PO 6 months; (6) PO 1 year; (7) PO 2 years.
Basic and instrumental Activities of Daily Living | Over 2 years
  This evaluation checklist will take under 5 minutes to assess participant's function status. Assessment to be performed at: (1) Baseline; (2) Postoperative(PO) day 14; (3) PO 6 week; (4) PO 3 months; (5) PO 6 months; (6) PO 1 year; (7) PO 2 years.
Basic Gait Assessment | Over 2 years
  Basic gait assessment will be performed including (A) Gait Speed, (B) Timed up and go test, (C) 5X sit to stand test. Assessment to be performed at: (1) Baseline; (2) Postoperative(PO) day 14; (3) PO 6 week; (4) PO 3 months; (5) PO 6 months; (6) PO 1 year; (7) PO 2 years.

SECONDARY OUTCOMES:
Fluid biomarkers | Over 1 year
  Blood plasma and cerebrospinal fluids will be analysed for biomarkers related to Alzheimer's disease, neurodegeneration and lymphatic dysfunction. Blood plasma will be sampled at (1) Operative day; (2) Postoperative(PO) day 3; (3) PO day 7; (4) PO day 14; (5) PO 6 weeks; (6) PO 3 months; (7) PO 6 months; (8) PO 1 year. CSF will be sampled at (1) Operative day; (2) PO day 7; (3) PO 6 weeks [Optional]; (4) PO 3 months [Optional].
Magnetic Resonance Imaging (MRI) of the Brain | Over 1 year
  Participants will undergo pre- and post-intervention MRI of the brain for evaluation of neuroanatomical pathology and surrogate markers of glymphatic function (eg. DTI-ALPS). The scans will be performed at (1) Baseline, (2) Postoperative Day 7, (3) Postoperative 3 months.
Positron Emission Tomography (PET) of the brain | Over 3 months
  Participants will undergo pre- and post-intervention PET fluorodeoxyglucose (FDG) brain scan to provide functional spatial information on changes before and after the surgery (at 3 months).

CONTACTS AND LOCATIONS:
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No